CLINICAL TRIAL: NCT03024424
Title: Value of Genetic Counseling and Testing for Patients Who Would Like to Know More About Their Personal Risk of AMD
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Utah (Other)
Responsible Party: Principal Investigator, Paul S. Bernstein, Professor, Ophthalmology/Visual Sciences, University of Utah
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: IRB 60413
Record Dates: First submitted 2017-01-11; First posted 2017-01-18 (Estimated); Last update posted 2023-05-06 (Actual); Status verified 2023-05

CONDITIONS: Age-Related Macular Degeneration; Choroidal Neovascularization; Genetic Counseling
MeSH Terms: conditions — Macular Degeneration; Choroidal Neovascularization

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Masking Description: Masking is applicable to risk of age-related macular degeneration, not to intervention assignment.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Early disclosure (Experimental): Early disclosure group receives results of genetic testing at Week 4
  Interventions: Behavioral: Early disclosure
- Late disclosure (Active Comparator): Late disclosure group receives results of genetic testing at final study visit (Month 12)
  Interventions: Behavioral: Late disclosure

INTERVENTIONS:
Behavioral: Early disclosure
  Arms: Early disclosure
Behavioral: Late disclosure
  Arms: Late disclosure

SUMMARY:
The goals of this study are:

To assess the impact of genetic testing based on how it alters behaviors, to assess the utility of serum biomarker measurement in combination with genetic testing, to assess the utility of genetic counseling in personal analysis of risk for age-related macular degeneration (AMD), and to assess the impact of presymptomatic genetic testing for choroidal neovascularization (CNV).

ELIGIBILITY:
Inclusion Criteria:

* Caucasian (this particular genetic test is only validated in Caucasians) Participants can have a positive family history of AMD but this is not necessary.

Exclusion Criteria:

* Individuals with a personal history of AMD are not eligible. Non-caucasian individuals are not eligible. Employees of the Moran Eye Center are not eligible.
* Individuals with a personal history of previous AMD genetic risk testing are not eligible.
* Individuals with a major psychiatric disorder

Ages: 18 Years to 64 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 16 (Actual)
Dates: Start 2016-03 (Actual); Primary Completion 2017-08-10 (Actual); Study Completion 2017-08-10 (Actual)

PRIMARY OUTCOMES:
Change in carotenoid levels in the skin | Twelve months
  Carotenoid levels in the skin are measured non-invasively at baseline and again at 12 months. Carotenoid levels are a biomarker of fruit and vegetable intake.
Change in carotenoid levels in the eyes | Twelve months
  Carotenoid levels in the eyes are measured non-invasively at baseline and again at 12 months.

CONTACTS AND LOCATIONS:
Overall Officials: Paul S. Bernstein, MD, PhD, Principal Investigator — University of Utah Moran Eye Center
Locations (1):
- University of Utah John A. Moran Eye Center, Salt Lake City, Utah, United States

IPD SHARING:
Plan to Share IPD: No